CLINICAL TRIAL: NCT00984152
Title: Open Label, Randomized Trial of TDF/FTC+Raltegravir Vs. TDF/FTC+Efavirenz in HIV-1-Infected Women: Differential Effects on Viral Suppression/Reservoir, & Immune Parameters in Different Compartments, Including Gut & Genital Tract
Brief Title: Trial of TDF/FTC + Raltegravir Versus TDF/FTC + Efavirenz in HIV-1-Infected Women
Acronym: ICE-002
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision not to go forth with study.
Sponsor: Rush University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Alan L. Landay, Ph.D., Rush University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08102303-IRB01; Merck IISP #33421
Record Dates: First submitted 2009-05-07; First posted 2009-09-25 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: HIV-1 Infections
Keywords: HIV; Raltegravir; Women; Viral Suppression; Viral Reservoir; Immune Parameters; Gut; Genital Tract
MeSH Terms: interventions — Raltegravir Potassium; efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): TDF/FTC Once-Daily + Raltegravir 400 mg Orally Twice-Daily
  Interventions: Drug: TDF/FTC Once-Daily + Raltegravir 400 mg Orally Twice-Daily
- 2 (Active Comparator): TDF/FTC + Efavirenz (Atripla) Once-Daily
  Interventions: Drug: TDF/FTC + Efavirenz (Atripla) Once-Daily

INTERVENTIONS:
Drug: TDF/FTC Once-Daily + Raltegravir 400 mg Orally Twice-Daily — TDF/FTC Once-Daily + Raltegravir 400 mg Orally Twice-Daily
  Other Names: TDF/FTC Once-Daily + Raltegravir (Isentress) 400 mg Orally Twice-Daily
  Arms: 1
Drug: TDF/FTC + Efavirenz (Atripla) Once-Daily — TDF/FTC + Efavirenz (Atripla) Once-Daily
  Arms: 2

SUMMARY:
Raltegravir not only has a unique mechanism of action, but may also have other unique effects on suppression of viral replication, viral reservoir, and immune reconstitution in blood and other important compartments. This may in part be due to the pharmacokinetics of Raltegravir in blood and gut tissue. Efavirenz will be the comparator antiretroviral drug in this study, with both drugs being used as part of a three-drug regimen with tenofovir and emtricitabine.

The primary objectives are to determine differences in the effects of 2 anti-retroviral regimens, Raltegravir + Truvada versus Atripla, with respect to:

1. Viral load in plasma, genital tract (vaginal secretions), and gut (by in situ hybridization).
2. Latent viral reservoir (pro-viral DNA) in the peripheral blood and genital tract.
3. Immune effects (CD4/CD8 immunophenotypes) in gut and PBMCs and plasma cytokine profiles.

The secondary objective is to determine the pharmacokinetics of Raltegravir in blood and gut tissue; relative tissue/compartment penetration compared to Efavirenz.

DETAILED DESCRIPTION:
This is a phase III, prospective, randomized (1:1), multicenter, open label study comparing the effects of two HAART regimens:

* Arm A: Raltegravir 400 mg PO BID + TDF/FTC (Truvada, 300/200 mg) One PO Daily
* Arm B: Efavirenz + TDF/FTC (Atripla) Once PO Daily

The following local sites: Mt. Sinai, Rush University Medical Center, Stroger Hospital, University of Chicago and University of Illinois will work together to enroll 10 eligible women meeting all eligibility criteria (5 per study arm) over a one year time period. These 10 women will be randomized 1:1 to receive either TDF/FTC + Raltegravir or TDF/FTC + Efavirenz (Atripla). There will be 2 baseline evaluations prior to initiation of study therapy. Subjects will be followed for 48 weeks after initiation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible subjects will be antiretroviral naïve (< 7 days of HAART at any time prior to entry) with plasma HIV-1 RNA > 50,000 copies/mL (obtained within 90 days prior to study entry by any laboratory that has a CLIA certification or its equivalent) and moderate immune suppression within 90 days prior to study entry.
2. HIV-1 infected, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test. Alternatively, if a licensed ELISA is not available, two HIV-1 RNA values >2000 copies/mL at least 24 hours apart performed by any laboratory that has CLIA certification or its equivalent may be used to document infection.
3. Female sex, Age > 18 and < 60 years, Pre-menopausal.
4. Screening CD4+ T-cell count between 200-350 cells/mm3 obtained within 90 days prior to study entry by any laboratory that has a CLIA certification or its equivalent.
5. The absence of exclusionary resistance mutations on a genotypic resistance assay (absence of exclusionary NRTI or NNRTI resistance mutations by genotype testing)
6. Antiretroviral (ARV) drug-naïve (defined as 7 days of ARV treatment at any time prior to entry).
7. Laboratory values obtained within 45 days prior to study entry:

   * Absolute neutrophil count (ANC) 500/mm3
   * Hemoglobin 8.0 g/dL
   * Platelet count 40,000/mm3
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase 5 ULN
   * Total bilirubin 2.5 x ULN
   * Calculated creatinine clearance ≥60 mL/min as estimated by the Cockcroft-Gault equation:

     * For women, multiply the result by 0.85 = CrCl (mL/min)
8. Negative serum or urine pregnancy test within 48 hours prior to initiating study medications unless otherwise specified by product labeling.

   * Female candidates of reproductive potential is defined as women who have had regular menses over the preceding 24 months
9. Contraception requirements for women who have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation).
10. Female candidates of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to the following:

    * If the regimen does not include EFV, they must agree to use at least one reliable method of contraception while receiving the protocol-specified drugs and for 6 weeks after stopping the medications.
    * If the regimen includes EFV, they must agree to use two reliable methods of contraception: a barrier method of contraception (e.g., condoms, diaphragm, or cervical cap with or without spermicide) together with another reliable form of contraceptive (e.g., a second barrier method, an IUD, or a hormone-based contraceptive) while receiving EFV and for 6 weeks after stopping EFV.

Exclusion Criteria:

1. Menopausal (may affect quantity of genital tract secretions) or any serious illness that requires treatment and/or hospitalization until the patient completes therapy
2. Any active infection, including co-infection with hepatitis B or C
3. Any neoplasm
4. Immunosuppressive therapy
5. Requirement for any medications that are prohibited by any of the study treatments
6. Significant liver or renal dysfunction
7. Baseline resistance to any of the study drugs by genotypic testing

   * NRTI: M41L, K65 R, D76N, T69D, K70R, L74V/I, y115F, Q151M, M184V, L210W, T215any, K219Q/E
   * NNRTI:L100I, K103N, V106A/M, V108I, Y181C/I, Y188C/L/H, G190anyA/S
8. Alcohol or substance abuse problems or psychiatric conditions that impair the ability of the subject to comply with the study protocol

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Viral load in plasma, genital tract (vaginal secretions), and gut (by in situ hybridization) | 48 weeks
Latent viral reservoir (pro-viral DNA) in the peripheral blood and genital tract | 48 weeks
Immune effects (CD4/CD8 immunophenotypes) in gut and PBMCs and plasma cytokine profiles | 48 weeks

SECONDARY OUTCOMES:
Determine the pharmacokinetics of Raltegravir in blood and gut tissue; relative tissue/compartment penetration compared to Efavirenz | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan L. Landay, Ph.D., Principal Investigator — Rush University Medical Center
Locations (5):
- United States (5):
  - Mt. Sinai Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - The Ruth M. Rothstein CORE Center (of Cook County), Chicago, Illinois
  - University of Chicago, Chicago, Illinois